CLINICAL TRIAL: NCT05229874
Title: A Prospective Randomized Controlled Study of the Efficacy of Carbon Nanoparticles Versus Indocyanine Green in Robotic or Laparoscopic Gastrectomy
Brief Title: Effect of CNSI vs. ICG in Lymph Node Tracing During Gastrectomy
Acronym: FUTURE-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUTURE-01
Record Dates: First submitted 2022-01-15; First posted 2022-02-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon nanoparticle suspension injection (CNSI) group (Experimental): CNSI (50 mg/dose) was produced by Chongqing Lesmei Pharmaceutical Co., Ltd.: Carbon nanoparticles were marked in the endoscopy division 1 day before surgery, and CNSI was injected submucosally at 4 points (proximal side, distal side, and left and right sides) 0.5-1 cm from the tumor edge under endoscopy. The test dose for each point was approximately 0.25 ml.
  Interventions: Drug: carbon nanoparticles
- Indocyanine green (ICG) group (Active Comparator): ICG (25 mg/dose) was produced by Dandong Yichuang Pharmaceutical. ICG was marked in the endoscopy division 1 day before surgery and injected submucosally at 4 points (proximal side, distal side, and left and right sides) 0.5-1 cm from the tumor edge under endoscopy. The test dose for each point was approximately 0.5 ml.
  Both procedures were performed by a designated medical practitioner.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: carbon nanoparticles — Endoscopic injection
  Other Names: carbon nanoparticle suspension injection
  Arms: Carbon nanoparticle suspension injection (CNSI) group
Drug: Indocyanine green — Endoscopic injection
  Other Names: ICG
  Arms: Indocyanine green (ICG) group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of carbon nanoparticle suspension injection and indocyanine green tracer-guided lymph node dissection during gastrectomy in patients with gastric cancer

DETAILED DESCRIPTION:
Da Vinci robot surgery XI system has fluorescence imaging function, which can realize indocyanine green lymph node tracking navigation technology in the operation. At the same time, the lymph node tracking effect of nano carbon suspension injection is not affected by equipment. The flexible mechanical arm of Da Vinci robot combined with the application of lymph node tracing technology makes the lymph node dissection of gastric cancer surgery more thorough, and also reduces the difficulty of surgery. Indocyanine green navigational lymphadenectomy can also be performed by fluorescence laparoscopy. By comparing the two tracer techniques, the lymph node tracer technique which is more suitable for robot or laparoscopic surgery system is selected to provide help and choice for clinical surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. clinical stage tumor 1-4a (cT1-4a), N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
4. No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations
5. Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
6. American Society of Anesthesiology score (ASA) class I, II, or III
7. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
4. History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
5. Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
6. History of other malignant disease within past five years
7. History of previous neoadjuvant chemotherapy or radiotherapy
8. History of unstable angina or myocardial infarction within past six months
9. History of cerebrovascular accident within past six months
10. History of continuous systematic administration of corticosteroids within one month
11. Requirement of simultaneous surgery for other disease
12. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
13. FEV1<50% of predicted values
14. Diffuse; widespread; plastica

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Total Number of Retrieved Lymph Nodes | 10 days
  Compare total number of retrieved lymph nodes in both group.

SECONDARY OUTCOMES:
The rate of black-stained/fluorescence | 10 days
  The number of black-stained/fluorescent lymph node in experimental group is divided by the total number of lymph nodes in active experimental group
Positive rate | 10 days
  The number of positive lymph nodes in black-stained/fluorescent lymph nodes is divided by the number of total black-stained/fluorescent lymph nodes in experimental group
False positive rate | 10 days
  The number of negative lymph nodes in black-stained/fluorescent lymph nodes is divided by the number of total black-stained/fluorescent lymph nodes in experimental group
Negative rate | 10 days
  The number of negative lymph nodes in not black-stained/fluorescent lymph nodes is divided by the number of total not black-stained/fluorescent lymph nodes in experimental group
False negative rate | 10 days
  The number of positive lymph nodes in not black-stained/fluorescent lymph nodes is divided by the number of total not black-stained/fluorescent lymph nodes in experimental group
Number of Metastasis Lymph Nodes | 10 days
  Compare number of positive lymph nodes in both group.
Morbidity and mortality rates | 30 days
  This is for the early postoperative complication and mortality, which defined as the event observed within 30 days after surgery.
3-year disease free survival rate | 36 months
  Disease-free survival is calculated from the day of surgery to the day of recurrence (When the specific date of recurrence of the tumor is unknown, the ending point is the date of death due to tumor causes). In the event that neither death nor recurrence of the tumor are observed, the end point is the final date that a patient is confirmed as relapse-free.
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Intraoperative blood loss | 1 day
  Intraoperative blood loss
Postoperative lymph node anatomy duration | 1 day
  Postoperative lymph node anatomy duration

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhao, Study Chair — Departments of Third Surgery, Fourth Hospital of Hebei Medical University
Locations (1):
- Fourth Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Tian Y, Pang Y, Yang P, Guo S, Ma W, Guo H, Liu Y, Zhang Z, Ding P, Zheng T, Li Y, Fan L, Zhang Z, Wang D, Zhao X, Tan B, Liu Y, Zhao Q. Effect of carbon nanoparticle suspension injection versus indocyanine green tracer in guiding lymph node dissection during radical gastrectomy (FUTURE-01): a randomized clinical trial. Int J Surg. 2025 Jan 1;111(1):609-616. doi: 10.1097/JS9.0000000000001873. PMID 38954670
- [Derived] Tian Y, Pang Y, Yang P, Guo H, Liu Y, Zhang Z, Ding P, Zheng T, Li Y, Fan L, Zhang Z, Zhao X, Tan B, Wang D, Zhao Q. The safety and efficacy of carbon nanoparticle suspension injection versus indocyanine green tracer-guided lymph node dissection during radical gastrectomy (FUTURE-01): A single-center randomized controlled trial protocol. Front Oncol. 2023 Jan 6;12:1044854. doi: 10.3389/fonc.2022.1044854. eCollection 2022. PMID 36686792